CLINICAL TRIAL: NCT03404076
Title: Optimized Response Assessment of Gastrointestinal Stromal Tumors Using Dual-Energy CT: Prospective Multicenter-Multinational Trial in Patients Undergoing Targeted Therapy With a TKI Inhibitor.
Brief Title: Unifying Advanced Treatment With Advanced Imaging
Acronym: GISTm3
Status: Completed | Type: Observational
Sponsor: Heidelberg University (Other)
Collaborators: Institute of Clinical Radiology and Nuclear Medicine Mannheim (Unknown); Siemens Healthcare Diagnostics Inc (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Peter Hohenberger, Prof. Dr. med., Heidelberg University
Other Study IDs: GIST m3
Record Dates: First submitted 2017-11-03; First posted 2018-01-19 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Gastrointestinal Stromal Tumor (GIST)
Keywords: Gastrointestinal Stromal Tumor (GIST); Dual Energy CT; Tyrosine Kinase Inhibitor (TKI)
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- GIST patients under TKI treatment: GIST patients under TKI treatment are subjected to Dual Energy CT
  Interventions: Diagnostic Test: Dual Energy CT

INTERVENTIONS:
Diagnostic Test: Dual Energy CT — Dual Energy CT is performed for diagnostic evaluation in gastrointestinal stromal tumor (GIST) patients undergoing tyrosine kinase inhibitor (TKI) treatment

SUMMARY:
The study investigates response assessment of gastrointestinal stromal tumors using Dual Energy CT (DECT) in patients undergoing targeted therapy with a TKI Inhibitor.

DETAILED DESCRIPTION:
Patients treated with targeted therapies by tyrosine kinase inhibition (TKI) almost always show different response patterns than tumors treated with cytotoxic chemotherapy. Tumor manifestations treated with targeted therapies often show only minor measurable changes in tumor size despite inhibition of tumor proliferation. Decrease in tumor size fulfilling the criteria of a partial remission according to RECIST may occur at a delayed stage of treatment after several months (PMID 19620483). Sometimes, even an initial increase of maximum tumor diameters may be observed although those patients are treatment responders with respect to 'hard' study endpoints like overall survival or progression free survival. As a result, patients often are misclassified too early as non-responders. As a consequence, successful treatment is not recognized or decisions towards a less effective second-line therapy are made.

Dual Energy CT (DECT) is a new and robust CT method that allows to exactly quantify the intra-tumoral amount of intravenously injected iodinated contrast material PMID 21822784). Thus, the technique can be considered as a simple and reliable surrogate of tumor Perfusion (PMID 21822784, 21934517, 20498609, 18677487). Initial studies have demonstrated a high accuracy of DECT in the differentiation of benign and malignant tumors in the kidney or lung (PMID 20498609, 18677487, 18796658). Furthermore, it has been demonstrated that the amount of iodine in lung tumors correlates with tumor glucose metabolism (PMID 21822784). These findings confirm the results of previous studies that have demonstrated the relationship between tumor perfusion, tumor microvessel density and glucose metabolism (PMID 15304661).

The hypothesis of the study is that DECT is the more accurate diagnostic tool to evaluate immediate therapeutic response in patients with GIST undergoing TKI inhibitor therapy (in most cases Glivec ®) than evaluating by RECIST, World Health Organization (WHO) and Choi criteria.

ELIGIBILITY:
Inclusion Criteria:

* General inclusion criteria for TKI treatment according to general medical standard procedures

Exclusion Criteria:

* General inclusion criteria for TKI treatment according to general medical standard procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: gastrointestinal stromal (GIST) patients under tyrosine kinase inhibitor (TKI) treatment
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival after a three year follow-up | 3 years follow up
  To visualize and to evaluate therapy response or stable disease of GIST patients undergoing TKI treatment by Dual Energy CT

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hohenberger, Prof., MD, Principal Investigator — Clinical for Surgery, Section SCOTCH
Locations (1):
- University Center Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Le Cesne A, Van Glabbeke M, Verweij J, Casali PG, Findlay M, Reichardt P, Issels R, Judson I, Schoffski P, Leyvraz S, Bui B, Hogendoorn PC, Sciot R, Blay JY. Absence of progression as assessed by response evaluation criteria in solid tumors predicts survival in advanced GI stromal tumors treated with imatinib mesylate: the intergroup EORTC-ISG-AGITG phase III trial. J Clin Oncol. 2009 Aug 20;27(24):3969-74. doi: 10.1200/JCO.2008.21.3330. Epub 2009 Jul 20. PMID 19620483
- [Background] Schmid-Bindert G, Henzler T, Chu TQ, Meyer M, Nance JW Jr, Schoepf UJ, Dinter DJ, Apfaltrer P, Krissak R, Manegold C, Schoenberg SO, Fink C. Functional imaging of lung cancer using dual energy CT: how does iodine related attenuation correlate with standardized uptake value of 18FDG-PET-CT? Eur Radiol. 2012 Jan;22(1):93-103. doi: 10.1007/s00330-011-2230-3. Epub 2011 Aug 7. PMID 21822784
- [Background] Apfaltrer P, Meyer M, Meier C, Henzler T, Barraza JM Jr, Dinter DJ, Hohenberger P, Schoepf UJ, Schoenberg SO, Fink C. Contrast-enhanced dual-energy CT of gastrointestinal stromal tumors: is iodine-related attenuation a potential indicator of tumor response? Invest Radiol. 2012 Jan;47(1):65-70. doi: 10.1097/RLI.0b013e31823003d2. PMID 21934517
- [Background] Graser A, Becker CR, Staehler M, Clevert DA, Macari M, Arndt N, Nikolaou K, Sommer W, Stief C, Reiser MF, Johnson TR. Single-phase dual-energy CT allows for characterization of renal masses as benign or malignant. Invest Radiol. 2010 Jul;45(7):399-405. doi: 10.1097/RLI.0b013e3181e33189. PMID 20498609
- [Background] Graser A, Johnson TR, Chandarana H, Macari M. Dual energy CT: preliminary observations and potential clinical applications in the abdomen. Eur Radiol. 2009 Jan;19(1):13-23. doi: 10.1007/s00330-008-1122-7. Epub 2008 Aug 2. PMID 18677487
- [Background] Chae EJ, Song JW, Seo JB, Krauss B, Jang YM, Song KS. Clinical utility of dual-energy CT in the evaluation of solitary pulmonary nodules: initial experience. Radiology. 2008 Nov;249(2):671-81. doi: 10.1148/radiol.2492071956. Epub 2008 Sep 16. PMID 18796658
- [Background] Yi CA, Lee KS, Kim EA, Han J, Kim H, Kwon OJ, Jeong YJ, Kim S. Solitary pulmonary nodules: dynamic enhanced multi-detector row CT study and comparison with vascular endothelial growth factor and microvessel density. Radiology. 2004 Oct;233(1):191-9. doi: 10.1148/radiol.2331031535. Epub 2004 Aug 10. PMID 15304661